CLINICAL TRIAL: NCT06722677
Title: A Multi-Center, Triple-Blind, Randomized, Sham-Controlled Trial Assessing the Efficacy and Safety of Rehabilitation Paired with Vagus Nerve Stimulation for Upper Extremity Motor Function in Patients with Ischemic Stroke (Repair Study)
Brief Title: A Trial of Rehabilitation Paired with VNS for Motor Function in Patients with Stroke (Repair Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G115R&PINS-C2-01-53
Record Dates: First submitted 2024-11-10; First posted 2024-12-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; Upper Extremity Paresis
Keywords: Stroke; Ischemic Stroke; Paresis; Upper Extremity Paresis; Vagus Nerve Stimulation; Neuromodulation; Randomized Controlled Trial; Rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Paresis; Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The device can be set as active VNS or sham VNS (the actual intensity is 0 mA). An unmasking programmer not involved in treatments or assessments will be messaged the group of the participant and set appropriate stimulation setting at baseline follow-up timepoint. Other masking researchers, including therapists and assessors, as well as the participant will not know the stimulation setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VNS group (Experimental): Active VNS paired with rehabilitation
  Interventions: Device: VNS; Other: Rehabilitation
- Control group (Active Comparator): Sham VNS paired with rehabilitation
  Interventions: Device: Sham VNS; Other: Rehabilitation

INTERVENTIONS:
Device: VNS — An neuromodulation treatment that delivers electrical impulses to the brain via the vagus nerve.
  Arms: VNS group
Device: Sham VNS — An neuromodulation treatment that delivers electrical impulses to the brain via the vagus nerve, the actual intensity is 0 mA.
  Arms: Control group
Other: Rehabilitation — Rehabilitation movements to improve upper limb function after stroke.

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of vagus nerve stimulation (VNS) paired with rehabilitation for enhancing upper extremity motor function after ischemic stroke.

Researchers will compare the outcomes of active VNS paired with rehabilitation against sham VNS (the actual intensity is 0 mA) also paired with rehabilitation, in order to assess improvements in arm motor function post-stroke.

Participants in this study will undergo a surgical procedure to implant the VNS system and will subsequently recieve a 6 weeks in-clinic therapy, followed by an additional 6 weeks home exercise. During the final 6 weeks, participants will either recieve in-clinic therapy or maintain their home exercise, depending on their assigned group.

DETAILED DESCRIPTION:
There are 6 follow-up timepoints in this trial:

1. Screening follow-up timepoint (V1): All participants will sign the informed consent form and receive pre-implant evaluation, including physical examination, brain magnetic resonance imaging, FMA-UE, WMFT, modified Ashworth sacle, BDI, ect.
2. Surgery follow-up timepoint (V2):All participants will be implanted with the VNS system, including the G115R IPG and L312 lead.
3. Baseline follow-up timepoint (V3): There is a baseline evaluation 7 to 14 days after the surgery, then participants will be randomly assigned to VNS group or Control group. The randomization will be stratified by baseline FMA-UE (20 to 35, 36 to 50), age (<50, ≥50) and research center (south centers, north centers).
4. Clinic rehabilitation follow-up timepoint (V4): Participants will receive standard clinic rehabilitation 3 days per week and lasting 6 weeks. Active VNS (VNS group) or sham VNS (Control group) will be paired with rehabilitation. Participants will be evaluated at the last day of this follow-up timepoint.
5. Home exercise follow-up timepoint (V5): Participants will take standard home exercise everyday in 6 weeks. Active VNS (VNS group) or sham VNS (Control group) will be paired with rehabilitation. At the last day, after evaluating, group assignment is unblinded.
6. Unmasking follow-up timepoint (V6): In this 6 weeks, all participants will receive active VNS. Participants in VNS group will still take standard home exercise, and participants in Control group will receive standard clinic rehabilitation again. Participants will be also evaluated at the last day of this follow-up timepoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22 years and <80 years, all gender is acceptable.
2. History of unilateral supratentorial ischemic stroke ≥ 9 months but < 10 years.
3. Upper Extremity motor section of the Fugl-Meyer Assessment score ≥20 and ≤50.
4. Right- or left-sided weakness of upper extremity.
5. Ability to communicate, understand, and give appropriate consent. Subjects can follow trial commands.
6. Subjects have good compliance and can complete the visits after surgery.

Exclusion Criteria:

1. History of hemorrhagic stroke.
2. Presence of ongoing dysphagia or aspiration difficulties.
3. Prior injury to vagus nerve, either bilateral or unilateral.
4. Subject receiving medication that may significantly interfere with actions of VNS on neurotransmitter systems at study entry, clinic rehabilitation follow-up timepoint, or home rehabilitation follow-up timepoint, such as centrally acting cholinoceptor blockers, centrally acting adrenoceptor blockers, norepinephrine re-uptake inhibitors, etc.
5. Botox injections within 4 weeks prior to enrollment through the unmasking follow-up timepoint (Visit 6).
6. Severe spasticity of the upper extremity (Modified Ashworth ≥ 3).
7. Significant sensory loss of the upper extremity (Upper Extremity sensory section of the Fugl-Meyer Assessment score < 6).
8. Severe depression (Beck Depression Scale > 29).
9. Current requirement, or likely future requirement, of diathermy.
10. Current use of any other stimulation device, such as a pacemaker or other neurostimulator.
11. Pregnancy or plans to become pregnant or to breastfeed during the study period.
12. Participated in any other clinical trials within the preceding 3 months.
13. Not considered to be applicable by the investigator.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Average Change | V4, 6 weeks after Baseline follow-up timepoint
  The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment). The FMA-UE will be analyzed for difference in average change at Clinic rehabilitation follow-up timepoint compared to Baseline follow-up timepoint (Difference in average change in FMA-UE from V3 to V4).

SECONDARY OUTCOMES:
Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Response | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint
  The Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Response is the percent of patients with a 6 point or greater improvement on the FMA-UE.
Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Average Change | V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).
Wolf Motor Function Test (WMFT) Average Change | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The Wolf Motor Function Test (WMFT) is an assessment scale of upper extremity functional level after stroke. The functional assessment range is an average of 15 sub-items with a range from 0 to 5, with 0 (meaning did not attempt) to 5 (meaning normal).
Wolf Motor Function Test (WMFT) Response | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint
  Wolf Motor Function Test (WMFT) Response is the percent of patients with a 0.4 point or greater improvement on the WMFT.
Beck Depression Inventory (BDI) Average Change | V6, 6 weeks after Home exercise follow-up timepoint
  The Beck Depression Inventory (BDI) is a self-report questionnaire used to identify overt behavioral characteristics of depression. Items are scored on a 4-point scale that ranges from 0 to 3. Ratings are summed to provide a total score ranging from 0 to 63.
Montreal Cognitive Assessment (MoCA) Average Change | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  MoCA is designed to assess cognitive function in patients. It assesses a number of different cognitive domains, including visuospatial and executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. The total score is 30, with higher scores indicating better cognitive function.
Motor Activity Log (MAL) Average Change | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The Motor Activity Log (MAL) consists of 30 activities of daily living such as using a towel, brushing teeth, and picking up a glass. The individual is asked to rate how often and how well each activity was performed with the more impaired arm. The response scale ranges from zero (never used) to 5 (same as pre-stroke)
Stroke impact scale (SIS) Average Change | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The Stroke Impact Scale (SIS) is a self-reported measure of stroke outcomes. Each item is selfrated on a 5-point Likert scale in terms of the difficulty the person has experienced in completing them after the score.
EQ-5D-3L Average Change | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The EQ-5D-3L is a general measure of health outcomes in any population. It is a self-report questionnaire which provides a simple descriptive profile and a single index value for health status.
Incidence of Adverse Events | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The incidence of adverse events occurred during the clinical trial, whether or not related to the device.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - The Xin Qiao Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Jiangbin Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Brain Hospital of Hunan Province The Second People's Hospital of Hunan Province, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing university Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

REFERENCES:
- [Background] Dawson J, Liu CY, Francisco GE, Cramer SC, Wolf SL, Dixit A, Alexander J, Ali R, Brown BL, Feng W, DeMark L, Hochberg LR, Kautz SA, Majid A, O'Dell MW, Pierce D, Prudente CN, Redgrave J, Turner DL, Engineer ND, Kimberley TJ. Vagus nerve stimulation paired with rehabilitation for upper limb motor function after ischaemic stroke (VNS-REHAB): a randomised, blinded, pivotal, device trial. Lancet. 2021 Apr 24;397(10284):1545-1553. doi: 10.1016/S0140-6736(21)00475-X. PMID 33894832
- [Background] Kimberley TJ, Prudente CN, Engineer ND, Pierce D, Tarver B, Cramer SC, Dickie DA, Dawson J. Study protocol for a pivotal randomised study assessing vagus nerve stimulation during rehabilitation for improved upper limb motor function after stroke. Eur Stroke J. 2019 Dec;4(4):363-377. doi: 10.1177/2396987319855306. Epub 2019 Jun 17. PMID 31903435
- [Background] Dawson J, Engineer ND, Prudente CN, Pierce D, Francisco G, Yozbatiran N, Tarver WB, Casavant R, Kline DK, Cramer SC, Van de Winckel A, Kimberley TJ. Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Stroke: One-Year Follow-up. Neurorehabil Neural Repair. 2020 Jul;34(7):609-615. doi: 10.1177/1545968320924361. Epub 2020 Jun 1. PMID 32476617
- [Background] Dickie DA, Kimberley TJ, Pierce D, Engineer N, Tarver WB, Dawson J. An Exploratory Study of Predictors of Response to Vagus Nerve Stimulation Paired with Upper-Limb Rehabilitation After Ischemic Stroke. Sci Rep. 2019 Nov 4;9(1):15902. doi: 10.1038/s41598-019-52092-x. PMID 31685853
- [Background] Dawson J, Engineer ND, Cramer SC, Wolf SL, Ali R, O'Dell MW, Pierce D, Prudente CN, Redgrave J, Feng W, Liu CY, Francisco GE, Brown BL, Dixit A, Alexander J, DeMark L, Krishna V, Kautz SA, Majid A, Tarver B, Turner DL, Kimberley TJ. Vagus Nerve Stimulation Paired With Rehabilitation for Upper Limb Motor Impairment and Function After Chronic Ischemic Stroke: Subgroup Analysis of the Randomized, Blinded, Pivotal, VNS-REHAB Device Trial. Neurorehabil Neural Repair. 2023 Jun;37(6):367-373. doi: 10.1177/15459683221129274. Epub 2022 Oct 13. PMID 36226541
- [Background] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257
- [Background] Hays SA, Khodaparast N, Hulsey DR, Ruiz A, Sloan AM, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation during rehabilitative training improves functional recovery after intracerebral hemorrhage. Stroke. 2014 Oct;45(10):3097-100. doi: 10.1161/STROKEAHA.114.006654. Epub 2014 Aug 21. PMID 25147331
- [Background] Hays SA, Khodaparast N, Sloan AM, Fayyaz T, Hulsey DR, Ruiz AD, Pantoja M, Kilgard MP, Rennaker RL 2nd. The bradykinesia assessment task: an automated method to measure forelimb speed in rodents. J Neurosci Methods. 2013 Mar 30;214(1):52-61. doi: 10.1016/j.jneumeth.2012.12.022. Epub 2013 Jan 23. PMID 23353133
- [Background] Khodaparast N, Kilgard MP, Casavant R, Ruiz A, Qureshi I, Ganzer PD, Rennaker RL 2nd, Hays SA. Vagus Nerve Stimulation During Rehabilitative Training Improves Forelimb Recovery After Chronic Ischemic Stroke in Rats. Neurorehabil Neural Repair. 2016 Aug;30(7):676-84. doi: 10.1177/1545968315616494. Epub 2015 Nov 4. PMID 26542082
- [Background] Khodaparast N, Hays SA, Sloan AM, Hulsey DR, Ruiz A, Pantoja M, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation during rehabilitative training improves forelimb strength following ischemic stroke. Neurobiol Dis. 2013 Dec;60:80-8. doi: 10.1016/j.nbd.2013.08.002. Epub 2013 Aug 15. PMID 23954448
- [Background] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving function and activities of daily living in patients after stroke. Cochrane Database Syst Rev. 2013 Nov 15;(11):CD009645. doi: 10.1002/14651858.CD009645.pub2. PMID 24234980
- [Background] Plow EB, Carey JR, Nudo RJ, Pascual-Leone A. Invasive cortical stimulation to promote recovery of function after stroke: a critical appraisal. Stroke. 2009 May;40(5):1926-31. doi: 10.1161/STROKEAHA.108.540823. Epub 2009 Apr 9. PMID 19359643
- [Background] Bolognini N, Pascual-Leone A, Fregni F. Using non-invasive brain stimulation to augment motor training-induced plasticity. J Neuroeng Rehabil. 2009 Mar 17;6:8. doi: 10.1186/1743-0003-6-8. PMID 19292910
- [Background] Adkins DL, Hsu JE, Jones TA. Motor cortical stimulation promotes synaptic plasticity and behavioral improvements following sensorimotor cortex lesions. Exp Neurol. 2008 Jul;212(1):14-28. doi: 10.1016/j.expneurol.2008.01.031. Epub 2008 Feb 20. PMID 18448100
- [Background] Barbay S, Nudo RJ. The effects of amphetamine on recovery of function in animal models of cerebral injury: a critical appraisal. NeuroRehabilitation. 2009;25(1):5-17. doi: 10.3233/NRE-2009-0495. PMID 19713615
- [Background] Walker-Batson D, Curtis S, Natarajan R, Ford J, Dronkers N, Salmeron E, Lai J, Unwin DH. A double-blind, placebo-controlled study of the use of amphetamine in the treatment of aphasia. Stroke. 2001 Sep;32(9):2093-8. doi: 10.1161/hs0901.095720. PMID 11546902
- [Background] Sawaki L, Butler AJ, Leng X, Wassenaar PA, Mohammad YM, Blanton S, Sathian K, Nichols-Larsen DS, Wolf SL, Good DC, Wittenberg GF. Constraint-induced movement therapy results in increased motor map area in subjects 3 to 9 months after stroke. Neurorehabil Neural Repair. 2008 Sep-Oct;22(5):505-13. doi: 10.1177/1545968308317531. PMID 18780885
- [Background] Takahashi CD, Der-Yeghiaian L, Le V, Motiwala RR, Cramer SC. Robot-based hand motor therapy after stroke. Brain. 2008 Feb;131(Pt 2):425-37. doi: 10.1093/brain/awm311. Epub 2007 Dec 20. PMID 18156154
- [Background] Zhang T, Zhao J, Li X, Bai Y, Wang B, Qu Y, Li B, Zhao S; Chinese Stroke Association Stroke Council Guideline Writing Committee. Chinese Stroke Association guidelines for clinical management of cerebrovascular disorders: executive summary and 2019 update of clinical management of stroke rehabilitation. Stroke Vasc Neurol. 2020 Sep;5(3):250-259. doi: 10.1136/svn-2019-000321. Epub 2020 Jun 28. PMID 32595138